CLINICAL TRIAL: NCT03640780
Title: Practical Pattern of Surgical Timing of Childhood Cataract in China
Status: Completed | Type: Observational
Sponsor: Sun Yat-sen University (Other)
Responsible Party: Principal Investigator, Haotian Lin, Prof., Sun Yat-sen University
Other Study IDs: CCPMOH2018- China8
Record Dates: First submitted 2018-08-18; First posted 2018-08-21 (Actual); Last update posted 2018-08-27 (Actual); Status verified 2018-08

CONDITIONS: Childhood Cataract
Keywords: surgical timing; cataract extraction; IOL implantation; childhood cataract; real-world data
MeSH Terms: interventions — Observation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- cataract extraction (CE): Patients received CE without IOL implantation in the first surgical stage, and received IOL implantation at secondary surgical stage.
  Interventions: Other: observation
- cataract extraction and IOL implantation: Patients received CE and IOL implantation in the first surgical stage.
  Interventions: Other: observation

INTERVENTIONS:
Other: observation — The surgical ages and other information between two groups were compared.

SUMMARY:
In the current study, the investigators analyzed the surgical RWD of 2,421 children with childhood cataracts from the Childhood Cataract Program of the Chinese Ministry of Health (CCPMOH) at the Zhognshan Ophthalmic Center and proposed data-based clinical experience for the timings of cataract extraction and IOL implantation.

ELIGIBILITY:
Inclusion Criteria:

* childhood cataracts present at the ZOC at the first time age: 0-18 years

Exclusion Criteria:

* complicated with other type of cataracts

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: hospital-based
Sampling Method: Non-Probability Sample
Enrollment: 2421 (Actual)
Dates: Start 2005-01 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Surgical age | 2005-2014
  the surgical ages of two groups

CONTACTS AND LOCATIONS:
Locations (1):
- Zhognshan Ophthalmic Center, Sun Yat-sen University, Guangzhou, Guangdong, China